CLINICAL TRIAL: NCT03319225
Title: A Study of the Distal Gut Microbiome and Its Relation to Gastrointestinal Transit After Spinal Cord Injury
Brief Title: Examining the Distal Gut Microbiome After Spinal Cord Injury
Status: Completed | Type: Observational
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Mark S. Nash, Ph.D., FACSM, Professor, University of Miami
Other Study IDs: 20170526
Record Dates: First submitted 2017-10-19; First posted 2017-10-24 (Actual); Last update posted 2018-10-09 (Actual); Status verified 2018-10

CONDITIONS: Spinal Cord Injury
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | US Export: No

GROUPS / COHORTS (3):
- Tetraplegia: Persons with Tetraplegia
- Paraplegia: Persons with Paraplegia
- Neurologically-intact: Neurologically-intact controls

SUMMARY:
The purpose of this research study is to learn more about the causes of gastrointestinal dysfunction after spinal cord injury. It has been thought that the microbiome (the community of bacteria in the body) may be one such cause. The study will examine whether changes in the distal gut microbiome are related to gastrointestinal dysfunction in persons with Spinal Cord Injury and Non-Disabled Controls.

ELIGIBILITY:
Persons with a Spinal Cord Injury:

Inclusion Criteria:

1. Age 18-65
2. ≥ 1 year post-injury
3. Spinal cord injury resulting in Tetraplegia or Paraplegia (C5-T6) and motor complete or incomplete (AIS A-C) impairment. Injury level and impairment will be confirmed by an American Spinal Injury Association (ASIA) exam conducted less than 2 years before study entry. If longer than 2 years, a certified rater will repeat the exam.
4. Self -reported history of constipation or other gastrointestinal dysfunction (e.g., extended bowel care time or difficulty in bowel emptying)
5. Willingness to participate in the study

Exclusion Criteria:

1. Currently hospitalized
2. American Spinal Injury Association (AIS) D-E
3. Self-reported history of Crohn's disease or diverticulitis, gastric blockage/obstruction or swallowing disorder
4. Gastrointestinal surgery ≤ 3 months prior to study
5. Implanted cardiac pacemaker, spinal cord stimulator, morphine (pain), or intrathecal pump
6. Concurrent use of surface functional electrical stimulation (FES)

Neurologically-Intact Persons:

Inclusion Criteria:

1. Age 18 or over
2. Willingness to participate in the study

Exclusion Criteria:

1. Self-reported history of Crohn's disease or diverticulitis, gastric blockage/obstruction or swallowing disorder
2. Gastrointestinal surgery ≤ 3 months prior to study
3. Implanted cardiac pacemaker, spinal cord stimulator, morphine (pain), or intrathecal pump

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Persons with a spinal cord injury; Neurologically-intact controls
Sampling Method: Non-Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2017-12-18 (Actual); Primary Completion 2018-01-09 (Actual); Study Completion 2018-01-09 (Actual)

PRIMARY OUTCOMES:
Characterize microbiome composition | Study day 7
  Characterize the distal gut microbiome within and across the three groups

SECONDARY OUTCOMES:
Gastrointestinal transit time | Study day 5
  Measured by "Smart Pill" wireless motility capsule during gastric emptying
Autonomic state | Baseline
  Autonomic tone will be assessed indirectly using heart rate variability by measuring the normal-to-normal QRS complexes of the PQRST waveform of the electrocardiogram (ECG)
Inflammatory state | Baseline
  Measured by protein levels of inflammatory biomarkers in plasma

CONTACTS AND LOCATIONS:
Overall Officials: Mark S Nash, Ph.D., Principal Investigator — University of Miami
Locations (1):
- University of Miami Miller School of Medicine, Miami, Florida, United States